CLINICAL TRIAL: NCT00164086
Title: Atorvastatin in Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bayside Health (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7/04
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2005-09

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — Atorvastatin

INTERVENTIONS:
Drug: atorvastatin

SUMMARY:
The purpose of this trial is to study the effects of a medication already widely used to treat cardiovascular disease and diabetes, in reducing the progression of myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Myeloma in remission

Exclusion Criteria:

* Adverse events (AEs) to statin, already on a statin, or contraindication to statin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Spencer, MBChB, FRACP, PhD, Principal Investigator — The Alfred
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia